CLINICAL TRIAL: NCT05852834
Title: Using YouTube to Learn Anatomy: Perspectives of Mexican Medical Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Raúl Sampieri Cabrera, Professor, Universidad Nacional Autonoma de Mexico
Other Study IDs: 052798S
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Learning Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed at exploring the popularity, impact, and usefulness of using YouTube in learning anatomy as perceived by Mexican medical students studying at different universities along the country

ELIGIBILITY:
Inclusion Criteria:

* Student of medicine

Exclusion Criteria:

* Not student of medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students of medicine in mexico
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
Use of Youtube | In the last year
  percentage of students that use youtube

CONTACTS AND LOCATIONS:
Locations (1):
- Ernesto Calderon, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided